CLINICAL TRIAL: NCT05241535
Title: A Phase 1, Randomized, Partial Double-Blind, Placebo- and Positive-Controlled, Three-way Crossover Study to Evaluate the Effect of MT-7117 on the QT/QTc Interval in Healthy Subjects
Brief Title: Study to Evaluate the Effect of a Single Oral Dose of MT-7117 on the QT/QTc Interval in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanabe Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: MT-7117-Z-103
Record Dates: First submitted 2022-01-06; First posted 2022-02-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Intervention Model Description: This is a Phase 1, randomized, partial double-blind, placebo and positive-controlled, three-way crossover study to evaluate the effect of a single oral dose of MT-7117, placebo, and positive control, moxifloxacin, on the QT/QTc interval in healthy subjects. The study consists of 3 treatments administered in a specific sequence as per the randomization list. Each subject will receive all 3 treatments over a specific sequence.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Partially blinded. Placebo tablets to match active MT-7117 tablets
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sequence 1 (starting with MT-7117 or Placebo) (Experimental): Treatment A or B (a single oral dose of MT-7117 or Placebo), Treatment C (a single oral dose of moxifloxacin)", then Treatment A or B (a single oral dose of placebo or MT-7117).
  Interventions: Drug: MT-7117; Drug: moxifloxacin; Drug: Placebo
- Sequence 2 (starting with MT-7117 or Placebo) (Experimental): Treatment A or B (a single oral dose of placebo or MT-7117), Treatment A or B (a single oral dose of MT-7117 or Placebo), then Treatment C (a single oral dose of moxifloxacin).
  Interventions: Drug: MT-7117; Drug: moxifloxacin; Drug: Placebo
- Sequence 3 (starting sequence with Moxifloxacin) (Experimental): Treatment C (A single oral dose of moxifloxacin), Treatment A or B (a single oral dose of placebo or MT-7117), then Treatment A or B (a single oral dose of MT-7117 or Placebo).
  Interventions: Drug: MT-7117; Drug: moxifloxacin; Drug: Placebo

INTERVENTIONS:
Drug: MT-7117 — oral
Drug: moxifloxacin — oral
Drug: Placebo — oral

SUMMARY:
The purpose of this study is to evaluate the effect of a single oral dose of MT-7117 on the QT/QTc interval in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent to participate in this study after reading the participant information sheet and Informed Consent Form (ICF) and having the opportunity to discuss the study with the Investigator or designee.
2. Healthy male or female subjects, 18-45 years of age, inclusive, at the time of signing the ICF.
3. Subjects must weigh at least 50 kilograms (kg) (110 pounds) but no more than 95 kg (209 pounds) and have a body mass index (BMI) 18.0 to 30.0 kg/m2 both inclusive at Screening and on Day -1.
4. Female subjects must not be lactating and must have a negative serum pregnancy test at screening and a negative urine pregnancy test within 24 hours before receiving the first dose of IMP (Investigational Medicinal Product).
5. Female subjects of childbearing potential and male subjects with a partner of childbearing potential must agree to use 2 effective methods of contraception (in female subjects, one method must be highly effective).
6. Male subjects must agree not to donate sperm and female subjects must agree not to donate ova until 3 months after the last dose of IMP.
7. In the Investigator's opinion, the subject can understand the nature of the study and any risks involved in participation and is willing to cooperate and comply with the protocol restrictions and requirements.

Exclusion Criteria:

1. Presence or history of any hepatobiliary disease at Screening, determined clinically significant by the Investigator after discussion with Sponsor's Responsible Physician. Current, or history of, clinically significant (in the opinion of the Investigator and Sponsor Responsible Physician) endocrine, respiratory, neurological, gastrointestinal, renal, cardiovascular disease, or history (within the last 2 years) of any clinically significant psychiatric/psychotic illness disorder (including anxiety, depression, and reactive depression).
2. Clinically relevant abnormal medical history, physical findings or laboratory values at Screening or Day -1 that could interfere with the objectives of the study or the safety of the subject, as judged by the Investigator.
3. Subject with a history of gastrointestinal surgery or disease known to affect absorption, metabolism, or excretion of the IMP (other than surgical history of appendectomy and hernia repair / herniorrhaphy / hernioplasty are permitted).
4. Subjects who have had major surgery within 3 months of Day 1.
5. Family history of long or short QT syndrome, hypokalemia, syncope, or Torsades de Pointes.
6. Clinically significant 12-lead ECG abnormalities, including subjects with QTcF of ≥450 msec at Screening or Day -1. A repeat assessment is allowed at each visit. If the repeat measurement is in range, the subject may be included.
7. Subjects with aspartate aminotransferase (AST), alanine aminotransferase (ALT), or bilirubin ≥1.5 × upper limit of normal reference range at Screening or Day -1. A repeat assessment is allowed at each visit. If the repeat measurement is in range, the subject may be included.
8. Blood pressure (supine) at Screening or Day -1 outside the range 90-145 mmHg (systolic) or 50-95 mmHg (diastolic); and resting heart rate (HR) outside the range of 45-100 bpm. A repeat assessment is allowed at each visit. If the repeat measurement is in range, the subject may be included.
9. Receipt of any prescribed or nonprescribed systemic or topical medication within 30 days (or, if relevant, 5 half-lives, whichever is longer) prior to the first dose of study drugs unless, in the opinion of the Investigator and Sponsor, the medication will not interfere with the study procedures or compromise subject safety.

   1. Occasional use of paracetamol (acetaminophen) for mild analgesia is permitted.
   2. Vitamins and herbal supplements are not permitted 14 days prior to dosing.
10. Presence or history of severe adverse reaction or allergy to any drug or excipient or other allergies that are of clinical significance to the study drugs.
11. Previously having received MT-7117.
12. History or presence of melanoma and/or lesions suspicious for melanoma at Screening.

    a. Subjects with the presence of a skin lesion suspicious for dysplastic nevus or a history of histologically proven dysplastic nevus.
13. Subjects with a first-degree relative with a history of familial melanoma.
14. Subjects who have previously received afamelanotide or melanotan.
15. Subjects who test positive for hepatitis B surface antigen, hepatitis B core antibody, hepatitis C antibody, or human immunodeficiency virus (HIV) 1 and HIV 2 antibodies at Screening.
16. Subjects who have had coronavirus disease 2019 (COVID-19) in the 3 months prior to Screening; or suspected active COVID-19 infection, a positive COVID-19 test, contact with an individual with known COVID-19, or travel to an area with a high risk of COVID-19 infection within 14 days of Screening or Day 1.

    1. Subjects who have received a COVID-19 vaccination within 14 days of Day 1. COVID-19 vaccination is not permitted during the study. Subjects may not take part in the study if they have started but not completed a COVID-19 vaccination course at the time of Screening or Day -1. Subjects who do not plan to complete the COVID-19 vaccination course will be allowed to participate in the study as long as at least 14 days have elapsed since the last vaccination.
    2. Subjects who test positive for COVID-19 at Day -1.
    3. Subjects currently suffering from clinically significant prolonged COVID symptoms.
17. Presence or history of drug abuse (as defined by Diagnostic and Statistical Manual of Mental Disorders [DSM-V] criteria), or a positive urine test for drugs of abuse at Screening or Day 1.
18. Presence or history (in the last 2 years) of alcohol abuse or excessive alcohol consumption, defined as subjects who regularly, or on average, drink more than 21 units (168 grams) for males or 14 units (112 grams) for females, of alcohol per week (1 unit is equivalent to 8 grams of alcohol).
19. Subjects who use tobacco or nicotine-containing products (snuff, chewing tobacco, cigarettes, cigars, pipes, e-cigarettes, or nicotine replacement products) within 3 months prior to dosing, or positive urine cotinine test at Screening or Day -1.
20. Consumption of food or drink containing licorice, oranges, or grapefruit from 7 days prior to dosing with IMP.
21. Subjects who are not willing to abstain from the consumption of caffeine and methylxanthine (e.g., coffee, tea, cola, energy drinks, or chocolates) in the 48 hours before Day -1 until completion of the post-treatment assessments on Day 2.
22. Donation of 1 or more units of blood (≥450 milliliters) in the 3 months prior to Screening, or plasma in the 7 days prior to Screening, or platelets in the 6 weeks prior to Screening, or intention to donate blood within 3 months after the last scheduled visit.
23. Heavy physical training, excessive exercise or heavy labor (e.g., long-distance running, weightlifting, or any physical activity to which the subject is not accustomed) from 3 days before the administration of the study drug.
24. Participation in any study* involving administration of an IMP within 8 weeks (or, if relevant, 5 half-lives, whichever is the longer) prior to the first dose. (*Disregarding any study Follow-up Periods).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-02-27 (Actual)

PRIMARY OUTCOMES:
Placebo-corrected, baseline-adjusted QTcF (corrected QT interval using the Fridericia formula) interval (ΔΔQTcF) at designed time points up to 24 hours post-dose | Pre-dose, 15 minutes post dose, 30 minutes post dose, 1 hour post dose, 2 hours post dose, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose
  The upper bound of the one-sided 95% confidence interval (CI) for the ΔΔQTcF at geometric mean Cmax (maximum plasma concentration) level is <10 milliseconds.

SECONDARY OUTCOMES:
Absolute values and changes in QTcF interval, PR (retrograde P waves), and QRS (Q wave, R wave, and S wave) values from Baseline at each timepoint. | Pre-dose, 15 minutes post dose, 30 minutes post dose, 1 hour post dose, 2 hours post dose, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose
Absolute values and changes in heart rate (HR) from Baseline at each timepoint. | Pre-dose, 15 minutes post dose, 30 minutes post dose, 1 hour post dose, 2 hours post dose, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose
The lower bound of the one-sided 95% CI of the ΔΔQTcF is >5 milliseconds at one or more individual timepoints between 1 hour and 4 hours after a single dose of moxifloxacin. | 1 hour post dose, 2 hours post dose, 3 hours post dose and 4 hours post dose
  Assay sensitivity.
The slope in concentration-response analysis for moxifloxacin is significantly positive from zero and the lower bound of the two-sided 90% CI of the predicted ΔΔQTcF at the geometric mean Cmax exceeds 5 milliseconds. | Pre-dose, 15 minutes post dose, 30 minutes post dose, 1 hour post dose, 2 hours post dose, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose
  Assay sensitivity.
Proportion of subjects with a QTcF interval >=450, >=480, and >=500 milliseconds. | Pre-dose, 15 minutes post dose, 30 minutes post dose, 1 hour post dose, 2 hours post dose, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose
Proportion of subjects with an increase from baseline in QTcF interval of >30 and >60 milliseconds. | Pre-dose, 15 minutes post dose, 30 minutes post dose, 1 hour post dose, 2 hours post dose, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose
Proportion of subjects with HR, PR interval, or QRS duration abnormalities. | Pre-dose, 15 minutes post dose, 30 minutes post dose, 1 hour post dose, 2 hours post dose, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose
  HR < 40 bpm (bits per minute) after a decrease of HR>=20 bpm from Baseline, or HR > 110 bpm after an increase of HR>=20 bpm from Baseline.
  PR interval of <100 milliseconds after a decrease of PR interval >= 25% from Baseline, or PR interval of >220 milliseconds after an increase of PR interval >= 25% from Baseline.
  QRS duration >120 milliseconds.
  Change of QRS duration >= 25% from baseline reaching a QRS >=120 milliseconds.
Proportion of subjects with an emergent ECG (Electrocardiogram) diagnostic abnormality. | Pre-dose, 15 minutes post dose, 30 minutes post dose, 1 hour post dose, 2 hours post dose, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose
Plasma concentration versus time profile of MT-7117 after dosing. | Pre-dose, 15 minutes post dose, 30 minutes post dose, 1 hour post dose, 2 hours post dose, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose
Plasma PK (Pharmacokinetics) parameters for MT-7117; maximum plasma concentration (Cmax) | Pre-dose, 15 minutes post dose, 30 minutes post dose, 1 hour post dose, 2 hours post dose, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose
Plasma PK parameters for MT-7117; time to maximum concentration (tmax) | Pre-dose, 15 minutes post dose, 30 minutes post dose, 1 hour post dose, 2 hours post dose, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose
Plasma PK parameters for MT-7117; area under the plasma concentration-time curve from zero to the last quantifiable concentration timepoint (AUC0-last) | Pre-dose, 15 minutes post dose, 30 minutes post dose, 1 hour post dose, 2 hours post dose, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose
Plasma PK parameters for MT-7117; area under the plasma concentration-time curve from zero to 24 hours (AUC0-24) | Pre-dose, 15 minutes post dose, 30 minutes post dose, 1 hour post dose, 2 hours post dose, 3, 4, 5, 6, 8, 10, 12, and 24 hours post-dose
Treatment-emergent AEs (Adverse Events) (including serious AEs [SAEs] and hepatic AEs of special interest [AESIs]). | Day-1 to Day 5 after Period 3.

CONTACTS AND LOCATIONS:
Overall Officials: Head of Medical Science, Study Director — Tanabe Pharma America, Inc.
Locations (2):
- United States (2):
  - Daytona Beach Clinical Research Unit, Daytona Beach, Florida
  - Dallas Clinical Research Unit, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No